CLINICAL TRIAL: NCT04774965
Title: The Effects of SlumberCurve™ Following Rotator Cuff Surgery: a Randomized Control Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to pursue study
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eight28, LLC (Unknown)
Responsible Party: Principal Investigator, Amit Momaya, Assistant Professor, Section Chief, Sports Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300006834
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tears; Surgery; Pain, Postoperative
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Slumber Curve Group (Experimental): Patients receiving Slumber Curve sleep aid for management of pain and sleep quality following rotator cuff repair.
  Interventions: Device: Slumber Curve sleep aid
- Normal Sleep Routine Group (No Intervention): Patients not receiving sleep aid.

INTERVENTIONS:
Device: Slumber Curve sleep aid — Patients who undergo rotator cuff repair and have been consented and randomized to the experimental group will be given a Slumber Curve sleep aid to be used during sleep. Each device will be numbered and recorded in the patient's REDCap entry for future reference if needed. Following administration of the Slumber Curve, patients will be given instructions on how to use the sleep aid while sleeping, and will be asked to use Slumber Curve nightly.
  Arms: Slumber Curve Group

SUMMARY:
The purpose of this study is to investigate the effects of a novel sleep aid known as SlumberCurve™, which serves as an adjustable form of a wedge pillow, on sleep quality and pain management following rotator cuff repair. The researchers hypothesize that SlumberCurve™ will significantly improve sleep quality and reduce night-time pain.

DETAILED DESCRIPTION:
Poor sleep quality is prevalent among patients undergoing rotator cuff repair surgery, and negatively affects the potential for proper healing. Without adequate sleep, the production of anabolic steroids and inflammatory cytokines are diminished. These anabolic steroids and inflammatory cytokines play a key role in postoperative healing, resulting in adequate pain regulation and increased patient satisfaction. Therefore adequate sleep quality is important not only for quality of life, but for postoperative healing. A recent systematic review revealed that some studies reported varying degrees in both the time and magnitude of change in return to adequate sleep quality following rotator cuff repair. This study hopes to address this gap in the literature by investigating a novel sleep aid, SlumberCurve, and its effect on sleep quality and night-time pain relief. SlumberCurve is a Class I Medical Device and is currently advocated to relieve tension and diminish pain in patients undergoing rotator cuff repair surgery. The device provides adjustable elevation of the torso as well as concave positioning, placing the shoulder in a more forward position. This novel sleep aid has the potential to increase sleep quality, and therefore enhance both patient satisfaction and postoperative recovery from rotator cuff repair surgery.

ELIGIBILITY:
Inclusion Criteria:

• Any male or nonpregnant female aged 18 years or older with a full-thickness rotator cuff tear undergoing rotator cuff repair surgery

Exclusion Criteria:

* Patients who receive workers' compensation benefits
* Patients with irreparable tears
* Patients undergoing revision surgery
* Patients with concomitant severe glenohumeral arthritis or concurrent adhesive capsulitis
* Sleep apnea disorder or other diagnosed sleep disorder
* Neuropsychiatric disease
* Use of sleep medication
* Prior shoulder surgery
* Rotator cuff arthropathy with pseudo paralysis
* Acute fractures involving the proximal humerus or shoulder girdle

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Fitbit Sleep Data - Time spent awake, restless, and asleep | 90 days
  Estimates of time spent awake, restless, and asleep will be assessed. All three measures will be recorded in minutes. Restless sleep indicates movement, and excessive movement will indicates time spent awake.
Fitbit Sleep Data - Sleep Stages | 90 days
  Sleep stages are estimated by utilizing movement and heart rate variability. Sleep stages are categorized into light sleep, deep sleep, and REM. Collective time spent in each stage will be recorded in minutes.
Pittsburgh Sleep Quality Index (PSQI) | 90 days
  The PSQI tracks sleep disturbances over time and includes seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleeping medications, and daytime dysfunction. Total of 21 points. Scores of less than 5 indicate adequate sleep. Scores of greater than 5 indicate poor sleep.
Visual Analog Scale (VAS) | 90 days
  Pain score, 0-10, 10 is best outcome
Single Assessment Numeric Evaluation (SANE) | 90 days
  Function score, 0-100%, 100% is best outcome
Postoperative Oral Morphine Equivalents | 90 days
  Oral morphine equivalents of all opioid-containing medications received
Simple Shoulder Test (SST) | 90 days
  Function score. Higher score indicates greater function.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kunze KN, Movasagghi K, Rossi DM, Polce EM, Cohn MR, Karhade AV, Chahla J. Systematic Review of Sleep Quality Before and After Arthroscopic Rotator Cuff Repair: Are Improvements Experienced and Maintained? Orthop J Sports Med. 2020 Dec 29;8(12):2325967120969224. doi: 10.1177/2325967120969224. eCollection 2020 Dec. PMID 33447619